CLINICAL TRIAL: NCT00387413
Title: A Double-blind, Double-dummy, Placebo-controlled, Incomplete Block, Two Period Crossover Study of the Histamine H3 Antagonist GSK189254 and Duloxetine in the Electrical Hyperalgesia Model of Central Sensitisation in Healthy Volunteers
Brief Title: A Study Of GSK189254 And Duloxetine In The Electrical Hyperalgesia Model Of Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: H3A106308
Record Dates: First submitted 2006-10-11; First posted 2006-10-13 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Hyperalgesia
Keywords: Duloxetine; GSK189254; Healthy volunteers; Phase I.; Electrical hyperalgesia model
MeSH Terms: conditions — Hyperalgesia | interventions — Duloxetine Hydrochloride; 6-((3-cyclobutyl-2,3,4,5-tetrahydro-1H-3-benzazepin-7-yl)oxy)-N-methyl-3-pyridinecarboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment Arm A1 (Experimental): In treatment Arm A1 Period 1 subject will receive 50 mcg GSK189254 plus Duloxetine Placebo in Week 1, in Week 2 subject will receive 100 mcg GSK189254 plus Duloxetine Placebo and in Week 3 subject will receive GSK189254 Placebo plus Duloxetine Placebo. In treatment Arm A1 Period 2 subject will receive GSK189254 Placebo plus Duloxetine Placebo for all 3 Weeks. There will be a washout of approximately one week between periods 1 and 2.
  Interventions: Drug: GSK189254; Drug: GSK189254 Placebo; Drug: Duloxetine Placebo
- Treatment Arm A2 (Experimental): In treatment Arm A2 Period 1 subject will receive GSK189254 Placebo plus Duloxetine Placebo for all 3 Weeks. In treatment Arm A2 Period 2 subject will receive 50 mcg GSK189254 plus Duloxetine Placebo in Week 1, in Week 2 subject will receive 100 mcg GSK189254 plus Duloxetine Placebo and in Week 3 subject will receive GSK189254 Placebo plus Duloxetine Placebo. There will be a washout of approximately one week between periods 1 and 2.
  Interventions: Drug: GSK189254; Drug: GSK189254 Placebo; Drug: Duloxetine Placebo
- Treatment Arm B1 (Experimental): In treatment Arm B1 Period 1 subject will receive 30 milligram (mg) Duloxetine plus GSK189254 Placebo in Week 1, in Week 2 60 mg Duloxetine plus GSK189254 Placebo and in Week 3 30 mg Duloxetine plus GSK189254 Placebo. In treatment Arm B1 Period 2 subject will receive GSK189254 Placebo plus Duloxetine Placebo for all 3 Weeks. There will be a washout of approximately one week between periods 1 and 2.
  Interventions: Drug: Duloxetine; Drug: GSK189254 Placebo; Drug: Duloxetine Placebo
- Treatment Arm B2 (Experimental): In treatment Arm B2 Period 1 subject will receive GSK189254 Placebo plus Duloxetine Placebo for all 3 Weeks. In treatment Arm B2 Period 2 subject will receive 30 milligram (mg) Duloxetine plus GSK189254 Placebo in Week 1, in Week 2 60 mg Duloxetine plus GSK189254 Placebo and in Week 3 30 mg Duloxetine plus GSK189254 Placebo. There will be a washout of approximately one week between periods 1 and 2.
  Interventions: Drug: Duloxetine; Drug: GSK189254 Placebo; Drug: Duloxetine Placebo

INTERVENTIONS:
Drug: Duloxetine — Subjects will be receive hard gelatin capsules of Duloxetine at 30mg once daily for one week and 60mg once daily for the second week in Treatment Arm B.
  Arms: Treatment Arm B1; Treatment Arm B2
Drug: GSK189254 — Subjects will receive film coated tablet of GSK189254 at 50 mcg once daily for a one week and 100 mcg once daily for the second week in Treatment Arm A.
  Other Names: Duloxetine
  Arms: Treatment Arm A1; Treatment Arm A2
Drug: GSK189254 Placebo — Subjects will receive Placebo matching GSK189254 for 3 weeks in each period.
Drug: Duloxetine Placebo — Subjects will receive Placebo matching Duloxetine for 3 weeks in each period.

SUMMARY:
GSK189254 is a highly potent histamine 3 (H3) receptor antagonist which has demonstrated efficacy in the reduction of mechanical hyperalgesia and allodynia in the chronic constriction injury pre-clinical model of neuropathic pain (NP). The mechanism of action of GSK 189254 in the pain model is hypothesised to be via enhanced release of monoamines in the central nervous system (CNS). A similar mechanism of action has also been shown for duloxetine. In this phase I study, the safety and efficacy of GSK189254 will be investigated in the electrical hyperalgesia (EH) model in healthy volunteers to build confidence that the preclinical efficacy demonstrated by this compound will translate into patients.

This study will be conducted as a double-blind, double-dummy, placebo-controlled, incomplete block, two period crossover study. Up to 40 healthy male or female volunteers, aged 18-45 years old, will be randomised into the study in order to achieve 32 evaluable subjects. Subjects will undergo two 3-week treatment periods and will be randomised to receive placebo and either GSK189254 (up to 100µg once daily) or duloxetine (up to 60mg daily). There will be a one week washout between treatment periods. The effects of repeated oral dosing of GSK189254 and duloxetine on secondary hyperalgesia in the EH model will be determined. Subject: GSK189254, Neuropathic pain (NP), H3 antagonist, duloxetine, Electrical hyperalgesia, Phase I, Healthy volunteers, Double blind, Safety, tolerability.

ELIGIBILITY:
Inclusion Criteria:

* He/she is a healthy subject.
* Women of child bearing potential must have a negative pregnancy test at screening and have undergone, or confirm regular use of one of the following:

Female sterilisation Sterilisation of male partner Practising a clinically accepted method of contraception during the study and for at least one month prior to baseline and one month following completion of the study.

* Has Caucasian skin colour.
* Body weight > 50kg and BMI within the range 18.5 to 29.9kg/m2 inclusive.
* Non smoker.
* Satisfactory pre-study medical within 28 days prior to the start of the study.
* No abnormality on clinical examination
* No abnormality on clinical chemistry or haematology.
* Negative pre-study urine drug screen and cotinine test.
* Signed and dated written informed consent prior to admission to the study.
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.
* Available to complete the study.

Exclusion Criteria:

* The subject has a positive pre-study urine drug/alcohol screen. A minimum list of drugs that will be screened for include Amphetamines, Barbiturates, Cocaine, Opiates, Cannabinoids, Methadone and Benzodiazepines.
* The subject has a history of drug or other allergy, that, in the opinion of the responsible physician, contraindicates their participation.
* A positive pre-study Hepatitis B surface antigen, positive Hepatitis C antibody or positive HIV results.
* History of clinically significant psychiatric disease, or presence of depressive disorder as defined by HAD depression score >8, or presence of anxiety disorder as defined by HAD anxiety score >8.

History or presence of insomnia or other sleep disorders.

* A QTcB interval < 430msec (men) or < 450msec (women).
* The subject has donated >500 mls of blood within 56 days prior to the first dose.
* Abuse of alcohol defined as an average daily intake of greater than 3 units for men and 2 units for the women.
* The subject has a history or presence of drug/substance abuse as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria.
* The subject has participated in a study with a new molecular entity during the previous 112 days or any other trial during the previous 84 days.
* The subject is currently taking regular (or a course of) medication whether prescribed or not. Such a subject may be included if the Investigator considers that this does not compromise safety or study procedures.
* Has received prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days or 5 half-lives whichever is the longer, prior to the first dose of study medication
* The subject has a history of chronic pain before screening.
* The subject has ingested or used a topical preparation containing aspirin or other non-steroidal anti-inflammatory drugs or paracetamol or other analgesic medication in the 7 days prior to the screening visit.
* The subject has used any topical steroid in the previous 30 days.
* The subject has used any topical capsaicin preparations on the forearms in the previous 30 days.
* The subject suffers from eczema, psoriasis or any other acute or chronic dermatological problem.
* The subject does not produce an area of allodynia or hyperalgesia to the EH model at screening
* The subject is unable to tolerate the EH model, including anxiety or atypical response to the model.
* The subject has any abnormality on diagnostic EEG at screening, or a history or presence of seizures or risk factors for seizure.
* The subject has any other medical condition that in the opinion of the Investigator would compromise the safety of the subject or the subject's ability to complete the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2006-10-02 (Actual); Primary Completion 2007-05-31 (Actual); Study Completion 2007-05-31 (Actual)

PRIMARY OUTCOMES:
Area of pin-prick hyperalgesia Area of touch-evoked allodynia | The mortality of above measurements at 7 months, functional status for each subject at 8-10 weeks.

SECONDARY OUTCOMES:
Ongoing pain intensity rating Area and intensity of flare Mood and alertness | The mortality for above measurements at 7 months, functional status for each subject 8-10 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- See also: Results for study H3A106308 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/H3A106308?search=study&search_terms=H3A106308#rs